CLINICAL TRIAL: NCT03776526
Title: Researching the Effects of Sleep on Step Count During the Postoperative Period Following Surgery for Hip Fracture
Brief Title: Researching the Effects of Sleep on STep Count dUring the Postoperative Period
Acronym: REST-UP
Status: Completed | Type: Observational
Sponsor: Christopher Patterson (Other)
Responsible Party: Sponsor-Investigator, Christopher Patterson, Professor Emeritus, McMaster University
Organization: McMaster University (Other)
Other Study IDs: REST-UP
Record Dates: First submitted 2018-07-26; First posted 2018-12-14 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Hip Fractures; Sleep; Postoperative Complications; Delirium
Keywords: Hip fractures
MeSH Terms: conditions — Hip Fractures; Postoperative Complications; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative Hip fracture patients: The target population will include patients aged 65 years or older admitted with hip fracture to the orthopedic ward at the Juravinski Hospital, a site of Hamilton Health Sciences Corporation in Ontario, Canada.
  Interventions: Behavioral: Fitbit® Alta HR Sleep monitoring

INTERVENTIONS:
Behavioral: Fitbit® Alta HR Sleep monitoring — Patients will be fitted with a Fitbit® Alta HR after surgery, which will monitor sleep quality (sleep duration and number of awakenings) for the duration of hospitalization.

SUMMARY:
Patients over the age of 65 who are admitted to the Juravinski Hospital for treatment of hip fractures will be invited to take part in the study. An activity monitor (a Fitbit® Alta HR) will be attached to the participant post-operatively, to record quality of sleep and amount of activity for the duration of hospital stay. The time spent in hospital and whether complications or confusion develops will also be recorded. The aim is to determine whether poor sleep affects recovery after hip fracture surgery.

DETAILED DESCRIPTION:
The purpose of this study is to examine the influence of sleep duration and quality on post-operative mobility in older adults admitted to hospital with a hip fracture. The hypothesis is that poor sleep will independently predict low post-operative mobility (measured by number of steps). Recent developments in activity monitor technology allow for the collection of reliable assessments of movement and sleep rhythm during surgical recovery.

The Fitbit® Alta HR activity monitor will be used for this study. When the participant is awake and alert after surgery and informed consent has been obtained, a study team member will fasten the Fitbit® device on the wrist of the participants' non-dominant hand. Investigators will monitor sleep quality and daily steps taken for the duration of hospitalization, with the option to discontinue if clinically required or requested by the patient or provider. At the time of discharge, the wearable biosensor will be reset and the information will be erased from its memory. The wearable biosensors will be cleaned with disinfectant used for durable medical equipment.

The study population will include patients aged 65+ admitted with hip fracture to the orthopedic ward (E2) at the Juravinski Hospital. Descriptive data on patients admitted with hip fracture will be collected including age, gender, Charlson comorbidity index, diagnosis of dementia, pre-hospital living accommodation, mobility aids, level of pre-admission mobility using the functional independence measure (FIM), and number of beds per room. Timing of surgery (within 24 hours, 48 hours, or more than 48 hours) after admission, highest reported daily pain score and foley catheter use will also be collected from the medical record. The use of sleep medications will be tracked each night during the study period. The physiotherapy notes will be screened for information on total distance ambulated in meters and in-hospital mobility progression. Post-operative complications such as Stroke, Cardiac event, Pneumonia, Venous thromboembolism, GI tract bleed, Urinary tract infections, Postoperative anemia, Acute Kidney Injury, and Pressure sores will be tracked from the medical record. Investigators will also contact participants by phone after 30 days have elapsed since discharge to inquire about mortality, FIM score and location of disposition.

The primary outcome is the total number of steps taken by participants during each 24-hour period after surgery for hip fracture. Mean daily steps will be calculated based on the number of days the activity monitor was worn. Secondary outcomes will be delirium prevalence, hospital length of stay, post-operative complications, 30-day post-discharge mortality, mobility status (FIM - locomotion subscale score), and location of disposition. The primary behavioural exposure is monitoring of sleep duration (measured by total sleep time in minutes) and quality (number of awakenings per night). Daytime naps will also be recorded.

One of the key strengths of this study is that both the primary outcome and the key exposure are measured using a single device, which improves the reliability and efficiency of data collection

ELIGIBILITY:
Inclusion Criteria:

* Patients recovering from surgery for hip fracture
* 65 years of age or older
* Able to provide informed consent or has a substitute decision maker able to provide consent

Exclusion Criteria:

* Bed or wheelchair bound prior to fracture
* Physical barrier to placement of device (wrist restraints, cast for wrist fracture)
* Non-operative hip fractures
* Pathologic hip fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to orthopedic ward after surgery for repair of hip fracture. Hamilton Health Sciences Corporation, Juravinski Hospital Site.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of steps per 24-hour day taken by patients during hospital admission after hip fracture repair. | Through study completion, on average 1 week
  Mean daily step count as measured by Fitbit®

SECONDARY OUTCOMES:
Delirium rate (incidence) | Through study completion, on average 1 week
  Delirium assessed by confusion assessment method (CAM)
Length of stay in hospital | Through study completion, on average 1 week
  Days from admission until discharge from hospital
Post-operative complications | Through study completion, on average 1 week
  Stroke, Cardiac event, Pneumonia, Venous thromboembolism, GI tract bleed, Urinary tract infections, Postoperative anemia, Acute Kidney Injury, and Pressure sores
30-day post-discharge mortality | 30 days post discharge
  Death within 30 days
30 day mobility status | 30 days post discharge
  Functional Independence Measure - locomotion subscale score
Location of disposition | Through study completion, on average 1 week
  community independent, community with home care, community with family support, inpatient rehabilitation, convalescent care, long term care, acute care hospital
Location of disposition at 30 days | 30 days post discharge
  community independent, community with home care, community with family support, inpatient rehabilitation, convalescent care, long term care, acute care hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided